CLINICAL TRIAL: NCT06240624
Title: Dynamic Brain Mapping of the Functional Effects of Levodopa on Multiple Cortex-basal Ganglia Circuits in Parkinson ́s Disease
Brief Title: Mapping Levodopa Effects on Cortico-basal Ganglia Circuit Function in Parkinson's Disease
Acronym: Dyn-fMRI-PD
Status: Active, not recruiting | Type: Observational
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-22010296
Record Dates: First submitted 2023-09-28; First posted 2024-02-05 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Levodopa-induced dyskinesia; Parkinson's disease; fMRI
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Parkinson's disease and Levodopa-induced dyskinesia: Inclusion criteria:
  * Aged 18 or more
  * Clinically established or probable PD according to the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's Disease
  * Peak-of-dose levodopa-induced dyskinesia
  * Stable antiparkinsonian medicine for 4 weeks
  * Signed informed consent
  Exclusion criteria:
  * Pregnancy or breastfeeding
  * History of other neurologic or psychiatric disease
  * Pacemaker or other implanted metallic or electronic devices which contraindicate MRI or TMS of the brain
  * Claustrophobia
  Interventions: Other: No intervention
- Patients with Parkinson's disease without Levodopa-induced dyskinesia: Inclusion criteria:
  * Aged 18 or more
  * Clinically established or probable PD according to the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's Disease
  * No levodopa-induced dyskinesia
  * Stable antiparkinsonian medicine for 4 weeks
  * Signed informed consent
  Exclusion criteria:
  * Pregnancy or breastfeeding
  * History of other neurologic or psychiatric disease
  * Pacemaker or other implanted metallic or electronic devices which contraindicate MRI or TMS of the brain
  * Claustrophobia
  Interventions: Other: No intervention
- Healthy controls: Inclusion criteria:
  * Aged 18 or more
  * Age- and sex-matched the PD groups
  * Signed informed consent
  Exclusion criteria:
  * Pregnancy or breastfeeding
  * History of other neurologic or psychiatric disease
  * Pacemaker or other implanted metallic or electronic devices which contraindicate MRI or TMS of the brain
  * Claustrophobia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be given.

SUMMARY:
Levodopa-induced dyskinesia (LID) in Parkinson's disease (PD) are involuntary movements caused by long-term treatment with dopaminergic replacement therapy (levodopa). During the cause of PD, most patients develop LID. In this study, the investigators plan to investigate how the cortico-basal-ganglia networks are affected in LID. The investigators will examine PD patients with and without LID as well as healthy age-matched controls using fMRI and PET. During the fMRI experiment, participants will perform a novel go-no task engaging both motor, emotional and reward brain networks. Patients will be scanned before and after intake of levodopa to study the dynamic effects of dopaminergic therapy. Furthermore, a dopamine transporter PET will be acquired to study the dopaminergic degeneration of the patients with PD.

DETAILED DESCRIPTION:
BACKGROUND Parkinson's disease (PD) is a neurodegenerative disease affecting the cortico-basal-ganglia network including dopaminergic degeneration. PD is treated with dopaminergic replacement therapy such as levodopa which is a natural precursor of dopamine. Unfortunately, most patients develop involuntary movements after many years of treatment which are called levodopa-induced dyskinesia (LID). Little is known about how brain networks are disturbed in LID. To investigate this, the investigators will conduct a multimodal characterization of PD patients with LID. Patients with and without LID will be studied using dynamic task-based fMRI to trace the levodopa-induced changes in functional brain activity and connectivity in the transition from the off-to-on medication state. For the task-based fMRI, the investigators will employ a novel experimental task that concurrently engages motor, emotional, and reward networks. Furthermore, the investigators will also map and quantify the dopaminergic presynaptic deficit using dopamine transporter (DAT) PET ([18F]PE2I-PET) to correlate the findings with MRI.

This study is part of a larger study of brain phenotyping PD (ADAPT-PD) with MRI.

AIM This sub-study aims to achieve a multimodal characterization of LID in PD using both fMRI and DAT PET. Furthermore, both motor, reward and emotional cortico-basal-ganglia networks will be investigated. The result of this study will lay the foundation of a future non-invasive brain stimulation study using transcranial magnetic stimulation (TMS) in PD.

HYPOTHESES

1. Patients with LID will show increased responsiveness to an acute levodopa challenge which will lead to a stronger time-dependent increase in striato-cortical motor network activity (preSMA and putamen) during NoGo trials after levodopa intake compared to patients without LID (Herz et al., 2014).
2. Patients with LID will show increased activity in the SMA and pre-SMA and less activity of the rIFG during movement (go responses) compared to patients without LID in the off-medication state (Cerasa et al., 2012).
3. Patients with LID will show abnormal levodopa-induced, task-related connectivity between putamen and and M1 compared to patients without LID (Herz et al., 2015).
4. Patients with LID will show decreased dopamine transporter activity in putamen compared to patients without LID (Hong et al. 2014).

The analysis regarding reward and emotional processing in patients with LID and the comparisons between fMRI and PET will be exploratory as no previous studies have been conducted.

RESEARCH PLAN For the sub-study, the investigators aim to recruit 25 PD patients with LID, 25 PD patients without LID, and 25 age-matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

• Aged 18 or more

Exclusion Criteria:

* Pregnancy or breastfeeding
* History of other neurologic or psychiatric disease
* History of epilepsy or familiar dispositions of epilepsy
* Pacemaker or other implanted metallic or electronic devices which contraindicate MRI or TMS of the brain
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, age- and sex-matched the PD groups
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Mean Change in Blood Oxygen-level Dependent (BOLD) Scores During Modified Go/No-Go Task | 4 task runs of 10 minutes each
  For each participant and each run, we will create general linear models with 20 regressors of interest.
  The regressors are Motor: Right, Left, and No-Go trials Emotion: Happy, Neutral, Sad Reward: High/low reward, high/low loss All above regressors will be separately modeled for the high- and the low-reward context.
  We will add a linear time modulation to all regressors to model dynamic changes in activation over time.
Peak force | 4 task runs of 10 minutes each
  Measured with grip-force response. The data will be smoothed and normalized to the individual maximum voluntary contraction.
Reaction time | 4 task runs of 10 minutes each
  Measured with grip-force response.
Maximum slope | 4 task runs of 10 minutes each
  Maximum value of first derivative of grip-force curve. Measured with grip-force response. The data will be smoothed and normalized to the individual maximum voluntary contraction.
Maximal negative slope | 4 task runs of 10 minutes each
  Maximum negative value of first derivative of grip-force curve. Measured with grip-force response. The data will be smoothed and normalized to the individual maximum voluntary contraction.
Parkinson's disease severity | Baseline (normal medication)
  Total Unified Parkinson's Disease Rating Scale (UPDRS) score (sum of all 4 subscores listed below, range 0-199, higher values = worse outcome), UPDRS-1 (Cognitive and mental disease severity, range 0-16, higher values = worse outcome), UPDRS-2 (disease severity in relation to activities of daily living, range 0-52, higher values = worse outcome) and UPDRS-3 (Motor severity, range 0-108, higher values = worse outcome), UPDRS-4 (Complications of therapy, range 0-23, higher values = worse outcome) subscores. Measured while subjects are taking their usual medication.
Motor disease severity | Before and 30-60 minutes after 150 % of normal morning levodopa dose as Madopar Quick.
  Unified Parkinson's Disease Rating Scale (UPDRS)-3 subscore (Motor severity, range 0-108, higher values = worse outcome). Measured while subjects are taking their usual medication.
  Unified Parkinson's Disease Rating Scale (UPDRS)-3 subscore (Motor severity, range 0-108, higher values = worse outcome). Measured while subjects are taking their usual medication.
  Unified Parkinson's Disease Rating Scale (UPDRS)-3 subscore (Motor severity, range 0-108, higher values = worse outcome). Measured while subjects are taking their usual medication.
Non-motor disease severity | Baseline
  Total Non-Motor Symptom Scale (NMSS) score (range 0-360, higher values = worse outcome). Measured while subjects are taking their usual medication.
Non-motor fluctuation severity | Baseline
  Total Non-Motor Fluctuation Assessment (NoMoFA) score (range 0-84, higher values = more severe non-motor fluctuations). Measured while subjects are taking their usual medication.
Modified Hoehn and Yahr Staging | Baseline
  Modified Hoehn and Yahr Staging (Crude measure of disease severity, range 0-5, higher score = worse outcome). Measured while subjects are taking their usual medication.
Schwab and England Activities of Daily Living Scale | Baseline
  Schwab and England Activities of Daily Living Scale (Measure of ADL function, range 100-0%, higher score = better ADL function). Measured while subjects are taking their usual medication.
Apathy | Baseline
  Total Lille Apathy Rating Scale (LARS) score (range -36-36, higher score = higher degree of apathy).
Depression | Baseline
  Major Depression Inventory (MDI) score (range 0-50), higher score = higher degree of depression
Impulsive-Compulsive Disorders (ICD) | Baseline
  Questionnaire for Impulsive-Compulsive Disorders (QUIP) (range 0-112), higher score = higher degree of ICD
Cognitive function | Baseline
  The Montreal Cognitive Assessment (MoCA) (range 0-30), higher score = better cognitive performance
Impulsivity | Baseline
  Barratt Impulsiveness Scale (BIS-11) (range 30-120), higher score = higher level of impulsivity.
Dyskinesia severity | Baseline (usual medication intake) as well as before and 30-60 minutes after 150 % of normal morning levodopa dose as Madopar Quick (range 0-104), higher score = higher dyskinesia severity
  Unified Dyskinesia Rating Scale (UDysRS)
Dopaminergic degeneration | Baseline
  Dopamine transporter (presynaptic) binding in the basal ganglia is measured using Fluorine-18 N-(3-iodopro-2E-enyl)-2beta-carbomethoxy-3beta-(4'-methylphenyl) nortropane Positron Emission Tomography to
Age | Baseline
Disease duration of Parkinson's disease | Baseline
Duration of levodopa-induced dyskinesia | Baseline
Medication | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Research Centre for Magnetic Resonance, Hvidovre Hospital, Hvidovre, Danmark, Denmark

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT06240624/Prot_SAP_ICF_000.pdf